CLINICAL TRIAL: NCT00028834
Title: A Phase II Trial Of Bevacizumab (NSC#704865) Plus Gemcitabine In Patients With Advanced Pancreatic Cancer
Brief Title: Bevacizumab and Gemcitabine in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02440; 11255B; N01CM17102 (NIH); CDR0000069138 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Bevacizumab

ARMS (1):
- Treatment (gemcitabine hydrochloride, bevacizumab) (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is to see if combining gemcitabine with bevacizumab works in treating patients who have advanced pancreatic cancer. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Combining chemotherapy with a monoclonal antibody may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate of patients with advanced pancreatic cancer who are treated with gemcitabine plus bevacizumab.

II. To determine the toxicity experienced by patients with advanced pancreatic cancer who are treated with gemcitabine plus bevacizumab.

III. To determine median and overall survival of patients with advanced pancreatic cancer who are treated with gemcitabine plus bevacizumab.

SECONDARY OBJECTIVES:

I. To measure plasma VEGF and serum VCAM-1 levels before, during, and after therapy as a predictor of outcome.

II. To collect and store serum samples for possible future assessment of other antiangiogenic inhibition markers.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * Not amenable to curative treatment with surgery or radiotherapy
  * Locally advanced disease must extend outside the boundaries of a standard radiation port
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Pleural effusions and ascites not considered measurable lesions
* No obvious tumor involvement of major vessels on CT scan
* No known brain metastases
* Performance status - ECOG 0-2
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No prior bleeding diathesis
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal
* PT INR no greater than 1.5
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* Urine protein less than 500 mg/24 hours if at least 1+ proteinuria
* No significant renal impairment
* No prior cardiovascular accident
* No prior deep vein thrombosis
* No myocardial ischemia or infarction within the past 6 months
* No uncompensated coronary artery disease within the past 6 months
* No uncontrolled hypertension
* No symptomatic congestive heart failure
* No cardiac arrhythmia
* No clinically significant peripheral artery disease
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction
* No prior pulmonary embolism
* No concurrent uncontrolled illness
* No ongoing or active infection
* No other concurrent active malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No psychiatric illness or social situation that would preclude study entry
* No prior allergic reaction attributed to compounds of similar chemical or biologic composition to bevacizumab or other agents (Chinese hamster ovary cell products or other recombinant human antibodies) used in this study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior bevacizumab
* No prior cytotoxic chemotherapy for metastatic disease
* No prior gemcitabine
* At least 4 weeks since prior adjuvant chemotherapy and recovered
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to sole site of measurable disease
* At least 6 weeks since prior major surgery
* At least 30 days since prior investigational agents
* At least 1 month since prior and no concurrent thrombolytic agents or full-dose anticoagulants (except to maintain patency of pre-existing permanent indwelling IV catheters)
* No concurrent chronic daily aspirin (more than 325 mg/day) or nonsteroidal anti-inflammatory drugs known to inhibit platelet function
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-02; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate (complete or partial responses) | Up to 2 years

SECONDARY OUTCOMES:
Progression-free survival | Up to 2 years
  Calculated using the Kaplan-Meier method, and the median progression-free survival times and the associated 95% confidence intervals derived.
Overall survival | Up to 2 years
  Calculated using the Kaplan-Meier method, and the median overall survival times and the associated 95% confidence intervals derived.

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States